CLINICAL TRIAL: NCT02058459
Title: A Sequential Two Phase Multicenter, Randomized Study to Optimize Dose Selection and Evaluate Safety After Treatment With the Holaira™ Lung Denervation System in Patients With Moderate to Severe COPD.
Brief Title: Targeted Lung Denervation for Patients With Moderate to Severe COPD
Acronym: AIRFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuvaira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AIRFLOW
Record Dates: First submitted 2014-02-05; First posted 2014-02-10 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Targeted Lung Denervation; Intervention; Lung Function; Safety; Device
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted Lung Denervation (Active Comparator): active targeted lung denervation
  Interventions: Device: Holaira™ Lung Denervation System with energy delivery
- Sham-Control (Sham Comparator): non-active targeted lung denervation
  Interventions: Device: Holaira™ Lung Denervation System without energy delivery

INTERVENTIONS:
Device: Holaira™ Lung Denervation System with energy delivery
  Arms: Targeted Lung Denervation
Device: Holaira™ Lung Denervation System without energy delivery
  Arms: Sham-Control

SUMMARY:
The purpose of this study is to evaluate safety of Targeted Lung Denervation (or TLD) in patients suffering from moderate to severe COPD. It is hypothesized that TLD will have a similar safety profile and improved physiological and functional outcomes to a sham-control.

DETAILED DESCRIPTION:
A prospective, sequential two phase multicenter, randomized double-blind, safety, & feasibility study. The goal of AIRFLOW-1 will be to compare two energy doses and select the optimal energy dose to be utilized in AIRFLOW-2. The goal of AIRFLOW-2 is to compare the optimal energy dose to a sham control. All subjects will be followed for a minimum of 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD with 30% ≤ FEV1 < 60% and FEV1/FVC <70% (post-bronchodilator);
* Patient ≥ 40 and ≤ 75 years of age at the time of consent;
* The patient has no child bearing potential or a negative pregnancy test (serum or urine), if applicable;
* Smoking history of at least 10 pack years;
* Non-smoking for a minimum of 2 months prior to consent and agrees to continue not smoking for the duration of the study;
* Participated in a pulmonary rehabilitation program or engaged in regular physical activity under professional supervision in the past 12 months;

Exclusion Criteria:

* Has been less than 6 weeks following the resolution of a COPD exacerbation or active lower respiratory infection (eg. pneumonia);
* History of recurrent respiratory infections and/or COPD exacerbations (more than 2 hospitalizations within 1 year of enrollment);
* Prior lung or chest procedure (eg. lung transplant, LVRS, BLVR, lung implant, metal stent, valves, coils, median sternotomy, bullectomy, segmentectomy, or lobectomy);
* Documented history of asthma diagnosed with onset <30 years of age, cystic fibrosis, paradoxical vocal cord motion, Churg-Strauss syndrome, allergic bronchopulmonary aspergillosis, severe interstitial lung disease or active tuberculosis;
* Pulmonary nodule requiring follow-up or intervention unless proven benign;
* Daily use of >10 mg of prednisone or its equivalent at the time of enrollment;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
AIRFLOW-1: Therapeutic interventions through 3 months; AIRFLOW-2: and rate of respiratory adverse events between 3 and 6.5 months | 3-6.5 months
  Respiratory adverse events is defined as: worsening bronchitis, worsening dyspnea, common cold, COPD exacerbation, influenza, pneumonia, respiratory infection, respiratory failure, tachypnea and wheezing. Subjects may have reported more than one type of respiratory adverse event.

SECONDARY OUTCOMES:
Adverse events over 3 years | 3 years
  The assessment of safety will be based on reporting of adverse events, particularly those adverse events that are respiratory in origin.
Device Success | 6 months
  Device success is defined as ability to deliver the test device to its intended locations, provide complete circumferential treatment and removal of the test device without the report of an adverse event during the procedure.
Spirometry measures | 3 years
  Measures include: FEV1, FVC, FEV1/FVC
Change in Functional testing: Cycle Ergometry & 6MWT | 3 years
Heath-related Quality of Life (SGRQ-C & EQ-5D) | 3 years
Procedure Success | Through discharge
  Procedure Success is defined as device success without the report of an adverse event through hospital discharge.
Plethysmography measures | 3 years
  Measures include Raw, TLC, IC, ITGW
CT Scan assessment | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD, Principal Investigator — University Medical Center Groningen; Arschang Valipour, MD, Principal Investigator — Otto-Wagner-Spital
Locations (18):
- Austria (2):
  - AKH Allgemeines Krankenhaus der Stadt Linz GmbH, Linz
  - Otto-Wagner-Spital, Vienna
- Belgium (2):
  - CHU Saint Pierre, Brussels
  - University Hospital Leuven, Leuven
- France (5):
  - CHU de Grenoble, Grenoble
  - CHU de Lille, Lille
  - CHU de Paris - Hopital Bichat Claude Bernard, Paris
  - CHU de Reims, Reims
  - CHU de Strasbourg, Strasbourg
- Germany (6):
  - Charite-Universitatsmedizin Berlin, Berlin
  - Universitatklinikum Bonn, Bonn
  - Ruhrlandklinik - West German Lung Center, Essen
  - Asklepios-Fachkliniken, Gauting
  - Thoraxklinik Heidelberg, Heidelberg
  - Klinikverbund Kempten-Oberallgaeu, Kempten
- Netherlands (2):
  - Universtity Medical Center Groningen, Groningen, The Netherlands
  - Academic Medical Center, Amsterdam
- Royal Brompton, London, United Kingdom

REFERENCES:
- [Derived] Valipour A, Shah PL, Herth FJ, Pison C, Schumann C, Hubner RH, Bonta PI, Kessler R, Gesierich W, Darwiche K, Lamprecht B, Perez T, Skowasch D, Deslee G, Marceau A, Sciurba FC, Gosens R, Hartman JE, Conway F, Duller M, Mayse M, Norman HS, Slebos DJ; AIRFLOW-2 Trial Study Group. Two-Year Outcomes for the Double-Blind, Randomized, Sham-Controlled Study of Targeted Lung Denervation in Patients with Moderate to Severe COPD: AIRFLOW-2. Int J Chron Obstruct Pulmon Dis. 2020 Nov 5;15:2807-2816. doi: 10.2147/COPD.S267409. eCollection 2020. PMID 33177818
- [Derived] Slebos DJ, Shah PL, Herth FJF, Pison C, Schumann C, Hubner RH, Bonta PI, Kessler R, Gesierich W, Darwiche K, Lamprecht B, Perez T, Skowasch D, Deslee G, Marceau A, Sciurba FC, Gosens R, Hartman JE, Srikanthan K, Duller M, Valipour A; AIRFLOW-2 Study Group. Safety and Adverse Events after Targeted Lung Denervation for Symptomatic Moderate to Severe Chronic Obstructive Pulmonary Disease (AIRFLOW). A Multicenter Randomized Controlled Clinical Trial. Am J Respir Crit Care Med. 2019 Dec 15;200(12):1477-1486. doi: 10.1164/rccm.201903-0624OC. PMID 31404499